CLINICAL TRIAL: NCT03438825
Title: The PREPARE-MVR Study: PRediction of Early PostoperAtive Right vEntricular Failure in Mitral Valve Replacement/Repair Patients
Brief Title: PRediction of Early PostoperAtive Right vEntricular Failure in Mitral Valve Replacement/Repair Patients
Acronym: PREPARE-MVR
Status: Completed | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: PREPARE-MVR1.0
Record Dates: First submitted 2018-02-11; First posted 2018-02-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Right Heart Failure; Right Ventricular Dysfunction; Right Ventricular Failure; Mitral Valve Disease
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Right | interventions — Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mitral valve replacement/repair — Mitral valve replacement/repair: standard of care operation of the mitral valve due to severe insufficiency

SUMMARY:
The PREPARE-MVR (PRediction of Early PostoperAtive Right vEntricular failure in Mitral Valve Replacement/Repair patients) Study aims to evaluate those preoperative factors which can predict the early postoperative right ventricular failure or determine the functional shift seen in right ventricular function after mitral valve replacement/repair. The PREPARE-MVR study focuses mainly on echocardiographic (both conventional and advanced) parameters and includes right heart catheterization intraoperatively and in the early postoperative period as gold standard method.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for mitral valve replacement/repair
* severe mitral valve insufficiency

Exclusion Criteria:

* preoperative right ventricular dysfunction
* cardiac surgery in medical history
* infective endocarditis
* primary cardiomyopathies
* congenital heart disease
* decreased left ventricular ejection fraction
* pulmonary embolism in medical history
* severe chronic obstructive pulmonary disease
* primary pulmonary hypertension
* any malignancy affecting right heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with isolated severe mitral valve insufficiency admitted for replacement/repair surgery as described in inclusion, exclusion criteria
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
right ventricular failure | From date of operation until the date of first documented right ventricular failure assessed up to 6 months
  Early postoperative right ventricular failure is defined as right ventricular stroke work index <300 mmHg/mL/m2 measured by right heart catheterization. Late right ventricular failure is defined as >10% decrease in right ventricular ejection fraction compared to preoperative value measured by 3D echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tokodi M, Nemeth E, Lakatos BK, Kispal E, Toser Z, Staub L, Racz K, Soltesz A, Szigeti S, Varga T, Gal J, Merkely B, Kovacs A. Right ventricular mechanical pattern in patients undergoing mitral valve surgery: a predictor of post-operative dysfunction? ESC Heart Fail. 2020 Jun;7(3):1246-1256. doi: 10.1002/ehf2.12682. Epub 2020 Mar 26. PMID 32220010